CLINICAL TRIAL: NCT02254265
Title: A Randomized, Multicenter, Double-Masked, Vehicle-Controlled, Dose-Ranging Study of the Safety and Efficacy of OTX-101 in the Treatment of Keratoconjunctivitis Sicca
Brief Title: Phase 2/3 Dose-Ranging Study of the Safety and Efficacy of OTX-101 in the Treatment of Keratoconjunctivitis Sicca
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OTX-101-2014-001
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Results first posted 2018-12-14 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2021-11

CONDITIONS: Keratoconjunctivitis Sicca; Dry Eye Disease
MeSH Terms: conditions — Keratoconjunctivitis Sicca; Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- OTX-101 0.05% (Experimental): OTX-101 0.05% ophthalmic solution 1 drop in both eyes BID for 84 days
  Interventions: Drug: OTX-101 0.05%
- OTX-101 0.09% (Experimental): OTX-101 0.09% ophthalmic solution 1 drop in both eyes BID for 84 days
  Interventions: Drug: OTX-101 0.09%
- Vehicle (Placebo Comparator): Vehicle of OTX-101 ophthalmic solution 1 drop in both eyes BID for 84 days
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: OTX-101 0.05% — OTX-101 0.05% Ophthalmic Solution
  Arms: OTX-101 0.05%
Drug: OTX-101 0.09% — OTX-101 0.09% Ophthalmic Solution
  Arms: OTX-101 0.09%
Drug: Vehicle — Vehicle of OTX-101 Ophthalmic Solution
  Arms: Vehicle

SUMMARY:
This is a Phase 2/3 study to evaluate the safety and efficacy of 2 different dose concentrations of OTX-101 dosed twice a day in both eyes for 84 days compared to placebo (vehicle) in patients with keratoconjunctivitis sicca (dry eye disease).

DETAILED DESCRIPTION:
Keratoconjunctivitis sicca (KCS) is a common multifactorial ophthalmologic disorder of the tears and ocular surface characterized by symptoms of burning, stinging, itching, grittiness, scratchiness, foreign body sensation, dryness, stickiness and tired eye sensation.

This study is the first clinical safety and efficacy study with OTX-101 and is designed to compare two dose concentrations of OTX-101 against vehicle (placebo) in reducing the signs and symptoms of KCS and evaluate safety when dosed twice a day in both eyes over an 84 day period.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age 18 years or older on the date of informed consent.
2. All subjects must provide signed written consent prior to participation in any study-related procedures.
3. Patient-reported history of KCS for a period of at least 6 months.
4. Clinical diagnosis of bilateral KCS supported by OTX-101-2014-001 study assessments.
5. Lissamine green conjunctival staining sum score of ≥ 3 to ≤ 9 out of a total possible score of 12 (scoring excludes superior zones 2 and 4) in the same eye at Screening and Baseline.
6. Global symptom score ≥ 40 at both Screening and Baseline.
7. Corrected Snellen VA of better than 20/200 in each eye.
8. Willing to discontinue use of current dry eye therapy (including artificial tears or ocular lubricants) during the study as of the run-in period.
9. Female subjects of childbearing potential must have a negative urine pregnancy test at Screening. Women of childbearing potential (ie, women who are not either postmenopausal for one year or surgically sterile) must use an acceptable form of contraception throughout the study.

Exclusion Criteria:

1. Use of cyclosporine ophthalmic emulsion 0.05% (Restasis®) within 3 months prior to Screening.
2. Previous treatment failure (lack of efficacy) on cyclosporine ophthalmic emulsion 0.05% (Restasis).
3. Diagnosed with Sjögren's disease ˃5 years prior to Screening.
4. Clinical diagnosis of seasonal and perennial allergic conjunctivitis.
5. Use of systemic and topical medications that are known to cause dry eye within 7 days prior to Screening and throughout the study period. These include the following medications:

   * Immunomodulators (permitted if dose is stable for 3 months prior to screening and does not change during the study period)
   * Antihistamines (including over-the counter (OTC))
   * Cholinergics
   * Antimuscarinics
   * Tricyclic antidepressants
   * Phenothiazines
   * Retinoids
6. Oral omega-3 fatty acids (permitted if dose is stable for 3 months prior to Screening and does not change during the study period)
7. Use of any topical ophthalmic medications, prescription (including antiglaucoma medications) or OTC (including artificial tears), other than the assigned study medication during the study period.
8. Current active eye disease other than KCS (i.e., any disease for which topical or systemic ophthalmic medication is necessary).
9. History of herpes keratitis.
10. Unstable macular disease (e.g., age-related macular degeneration, diabetic maculopathy). Stable macular disease is defined as no reduction in central VA within 6 months prior to Screening.
11. Diagnosis of chronic uveitis.
12. Corneal transplant (e.g., penetrating keratoplasty, lamellar keratoplasty, Descemet's stripping endothelial keratoplasty (DSEK) ).
13. Corneal refractive surgery (e.g., laser-assisted in situ keratomileusis (LASIK]) photo refractive keratectomy (PRK), limbal relaxing incision (LRI) ) within 6 months prior to screening or postoperative refractive surgery symptoms of dryness that have not resolved.
14. Cataract surgery within 3 months prior to Screening.
15. Non-laser glaucoma surgery at any time; glaucoma laser procedures within 3 months prior to Screening.
16. Presence of punctal plugs or past history of permanent punctal occlusion (e.g., cautery).
17. Lagophthalmos or clinically significant eyelid margin irregularity of the study eye whether congenital or acquired.
18. Presence of conjunctivochalasis (i.e., mechanical blockage of the lower lid punctum by redundant conjunctiva).
19. Presence of pterygium in the study eye.
20. Unwilling to discontinue use of contact lenses during the duration of the study.
21. Preplanned elective surgery or hospitalization during the study period.
22. HIV-positive.
23. Unable to reliably report symptoms and history.
24. Has known hypersensitivity or contraindication to the study medication(s) or their components.
25. Has a history or presence of chronic generalized systemic disease that the Investigator feels might increase the risk to the subject or confound the result(s) of the study.
26. Has a severe/serious ocular condition, or any other unstable medical condition that, in the Investigator's opinion, may preclude study treatment or follow-up.
27. Women who are pregnant or breastfeeding.
28. Participation in any drug or device clinical investigation within 30 days prior to entry into this study and/or during the period of study participation.
29. Previous randomization into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OTX-101 0.05% | OTX-101 0.09% | Vehicle
Started | 151 | 152 | 152
Completed | 142 | 140 | 144
Not Completed | 9 | 12 | 8

BASELINE CHARACTERISTICS:
Population: Intent to treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | OTX-101 0.05% | OTX-101 0.09% | Vehicle | Total
Number analyzed (Participants) | 151 | 152 | 152 | 455
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (13.27) | 59.2 (14.55) | 59.3 (13.75) | 60.1 (13.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 122 | 120 | 361
  Male | 32 | 30 | 32 | 94
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 8 | 7 | 3 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 2 | 2
  Black or African American | 11 | 13 | 20 | 44
  White | 128 | 126 | 120 | 374
  More than one race | 3 | 6 | 7 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Conjunctival Staining
Description: Mean change from baseline at day 84 for the lissamine green conjunctival staining score in the designated study eye.
  The Investigator recorded a score for each area of each eye on a 0 (No punctate stain in zone) to 3 (Densely concentrated micropunctate stain spots) scale
Time Frame: Baseline to 84 days
Population: Intent to treat population, last observed carried forward approach
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OTX-101 0.05% | OTX-101 0.09% | Vehicle
Number analyzed (Participants) | 151 | 152 | 152
score on a scale | -1.9 (2.17) | -1.8 (2.27) | -1.2 (2.17)

2. Primary Outcome: Global Symptom Score
Description: Mean change from baseline at day 84 for the global symptom score.
  The freuency and severy of dry eye and irritation scores were used to calculate symptom score as follows:
  Frequency of dry eye/irritation based on a scale of 0 (rarely) to 100 (all the time) Severity of dryness or irritation based on a scale of 0 (very mildly) to 100 (very severe).
  The global symptom score was calculated as the square root of the frequency score times the severity score
Time Frame: Baseline to 84 days
Population: Intent to treat population, observed data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OTX-101 0.05% | OTX-101 0.09% | Vehicle
Number analyzed (Participants) | 143 | 140 | 144
score on a scale | -19.78 (23.791) | -18.86 (22.810) | -19.16 (22.973)

3. Secondary Outcome: Tear Film Break up Time (TBUT)
Description: Mean change from baseline in TBUT in the study eye from baseline at Day 84
Time Frame: Baseline to 84 days
Population: Intent to treat population - observed data
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | OTX-101 0.05% | OTX-101 0.09% | Vehicle
Number analyzed (Participants) | 143 | 140 | 144
seconds | 0.43 (2.032) | 0.53 (2.590) | 0.39 (2.149)

4. Secondary Outcome: Corneal Staining Score
Description: Mean Change from Baseline in Corneal Staining Score in the Study Eye. Expanded National Eye Institute Scale for Corneal Staining Score was used to grade each of the 5 areas of the cornea on a 0 (No punctate stain in area) to 4 (Severe diffuse (coalescent) macropunctate stain of the area) scale
Time Frame: Baseline to 84 days
Population: Intent to treat population, Last observed carried forward approach
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OTX-101 0.05% | OTX-101 0.09% | Vehicle
Number analyzed (Participants) | 151 | 152 | 152
score on a scale | -1.4 (3.23) | -1.4 (2.87) | -0.6 (2.76)

5. Secondary Outcome: Schirmer's Test
Description: Change from Baseline in Categorized Schirmer's Test Score. Schirmer's test was performed with strips placed in both eyes at the same time. Strips were removed after 5 minutes and the amount of wetting (in mm) was recorded as scores from 1 to 5.
  1: < 3 mm, 3 - 6 mm, 7 - 10 mm, 11 - 14 mm, and 5: > 14 mm
Time Frame: Baseline to 84 days
Population: Intent to treat population (with both eyes averaged)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OTX-101 0.05% | OTX-101 0.09% | Vehicle
Number analyzed (Participants) | 143 | 140 | 144
score on a scale | 0.41 (1.263) | 0.37 (1.260) | -0.08 (1.307)

6. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction with treatment score using 5-point scale (1=extremely dissatisfied to 5=extremely satisfied)
Time Frame: Baseline to 84 days
Population: Intent to treat population (Observed)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OTX-101 0.05% | OTX-101 0.09% | Vehicle
Number analyzed (Participants) | 143 | 140 | 144
score on a scale | 3.8 (1.17) | 3.7 (1.17) | 3.9 (1.08)

ADVERSE EVENTS:
Arm/Group | OTX-101 0.09% | OTX-101 0.05% | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/152 | 0/151 | 0/152
Serious Adverse Events (participants affected / at risk) | 1/152 | 0/151 | 4/152
Other Adverse Events (participants affected / at risk) | 37/151 | 31/152 | 30/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OTX-101 0.09% (N=152) | OTX-101 0.05% (N=151) | Vehicle (N=152)
Peripheral nerve decompression (Surgical and medical procedures) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OTX-101 0.09% (N=151) | OTX-101 0.05% (N=152) | Vehicle (N=152)
Eye irritation (Eye disorders) | 3 | 2 | 1
Lacrimation increased (Eye disorders) | 3 | 2 | 1
Meibomian gland dysfunction (Eye disorders) | 2 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 1 | 2 | 2
Eye discharge (Eye disorders) | 1 | 2 | 0
Eye pruritus (Eye disorders) | 1 | 3 | 4
Vitreous floaters (Eye disorders) | 1 | 1 | 2
Eye pain (Eye disorders) | 0 | 0 | 2
Eyelid pain (Eye disorders) | 0 | 2 | 0
Vision blurred (Eye disorders) | 0 | 1 | 4
Vitreous detachment (Eye disorders) | 0 | 3 | 0
Instillation site pain (General disorders) | 23 | 20 | 5
Instillation site reaction (General disorders) | 0 | 2 | 1
Conjunctivitis viral (Infections and infestations) | 0 | 0 | 2
Corneal abrasion (Eye disorders) | 0 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 3 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2
Tremor (Nervous system disorders) | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Nasopharyngitis (Infections and infestations) | 2 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes